CLINICAL TRIAL: NCT04980716
Title: Early Specialized Cardiovascular Intervention Based on Impedance Cardiography in Locally Advanced Non-small Cell Lung Cancer Patients Who Receiving Radical Concurrent Chemoradiotherapy and Immunotherapy: a Prospective, Randomized Controlled, Multicenter Phase III Clinical Trial.
Brief Title: Early Specialized Cardiovascular Intervention Based on Impedance Cardiography in Locally Advanced Non-small Cell Lung Cancer Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-1074
Record Dates: First submitted 2021-07-24; First posted 2021-07-28 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Non-small Cell Lung Cancer; Cardiovascular Complication
Keywords: Non-small Cell Lung Cancer; Cardiovascular Intervention; Impedance Cardiography; Cardiovascular Event
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The early intervention group (Experimental): The early intervention group: evaluation and intervention based on impedance cardiography results at multiple timepoints. Specific intervention measures include:
  1. cardiovascular drug treatment: based on the increase and decrease of the "Golden Triangle"
     1. ACEI, perindopril tert-butyrate 4mg qd
     2. β receptor antagonist, metoprolol succinate 47.5mg qd
     3. Spironolactone 20mg qd
     4. Drugs to improve myocardial metabolism: trimetazidine hydrochloride 35 mg bid
     5. Other therapeutic drugs include: loop diuretics, ARNI, sinus node If current selection specific inhibitors, statins, antiplatelet aggregation and nitrate drugs, etc.
  2. Exercise intervention: exercise prescription based on the initial cardiopulmonary exercise test results.
  Interventions: Drug: Multiple cardiovascular drugs related to "Golden Triangle"
- The control group (No Intervention): This group will be under observation. When cardiovascular events (including ischemic cardiomyopathy, heart failure, arrhythmia requiring treatment, pericardial disease requiring treatment, valvular disease, etc.) happen, a cardiovascular specialist assessment and intervention will be given.

INTERVENTIONS:
Drug: Multiple cardiovascular drugs related to "Golden Triangle" — Based on impedance cardiography results at each timepoints, cardiovascular drug treatment and exercise plan will be given in the intervention group.
  Arms: The early intervention group

SUMMARY:
This is a prospective, randomized, controlled, multi-center phase III clinical trial that intends to evaluate the role of early cardiovascular intervention based on impedance cardiography in patients with locally advanced non-small cell lung cancer receiving radical radiochemotherapy±immunotherapy.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, multi-center phase III clinical trial that intends to evaluate the role of early cardiovascular intervention based on impedance cardiography in patients with locally advanced non-small cell lung cancer receiving radical radiochemotherapy±immunotherapy. The participants were 1:1 randomized to the intervention group and the control group. The intervention group will receive cardiovascular evaluation and intervention at multiple timepoints throughout treatment and follow-up, while the control group will be under observation unless severe cardiovascular events happen.

The evaluation and intervention timepoints include: Before neoadjuvant therapy, before radiotherapy, Mid-radiotherapy, 2 months after the completion of radiotherapy, every 6 months thereafter for up to 2 years post-radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. It is diagnosed as non-small cell lung cancer by pathological examination or cytological examination; it is assessed as locally advanced, unresectable stage III non-small cell lung cancer by imaging;
2. Plan to receive radical radiotherapy and chemotherapy ± immunotherapy;
3. Male or female between 18 and 75 years old;
4. Life expectancy ≥ 12 weeks;
5. The World Health Organization (WHO) PS score is 0 or 1;
6. Organ and bone marrow function meet the following conditions: Forced expiratory volume per second (FEV1) ≥1000 ml; absolute neutrophil count ≥1.5×10^9/L; platelets ≥100×10^9/L; hemoglobin ≥90 g/L ; Serum creatinine clearance calculated according to the Cockcroft-Gault formula ≥50 mL/min (Cockcroft and Gault 1976); serum bilirubin ≤1.5 times the upper limit of normal (ULN); alanine aminotransferase and aspartate aminotransferase ≤2.5 times ULN;
7. A signed informed consent form is required before proceeding with any step in the research;
8. There is an abnormality in the initial cardiac output index.

Exclusion Criteria:

1. PS score 2-4;
2. Organ function impairment: FEV1 <1000ml; absolute neutrophil count <1.5×10^9/L; platelets <100×10^9/L; hemoglobin <90 g/ L; Serum creatinine clearance calculated according to Cockcroft-Gault formula <50 mL/min; serum bilirubin>1.5 times ULN; alanine aminotransferase and aspartate aminotransferase>2.5 times ULN;
3. Unstable angina or myocardial infarction occurred in the past month;
4. Arrhythmia that has not been controlled and can cause symptoms or abnormal hemodynamics;
5. Active endocarditis;
6. Symptomatic severe aortic stenosis;
7. Heart failure that has not been controlled;
8. Acute pulmonary embolism, pulmonary infarction or low thrombosis (artery or vein) formation;
9. Suspected or confirmed aortic dissection;
10. Uncontrolled bronchial asthma;
11. Pulmonary edema;
12. Fingertip blood oxygen saturation at rest ≤85%;
13. Acute non-cardiopulmonary diseases (such as infection, renal failure, thyrotoxicosis, etc.) that may affect sports performance or aggravate due to exercise;
14. Mental disorders make it impossible to cooperate.
15. Patients for whom drug intervention is clearly recommended according to the 2022 edition of the European Society of Cardiology Guidelines on Cardio-Oncology.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2-year
  It was calculated from the first day of treatment to the day of death.
The incidence of grade 2+ cardiotoxicity events | 2-year
  Culmulative incidence of grade 2+ cardiotoxicity events

SECONDARY OUTCOMES:
Progression-free survival | 2-year
  From the first day of treatment to the day of progression or the day of death.
The incidence of grade 2+ pulmonary toxicity | 2-year
  Culmulative incidence of grade 2+ pulmonary toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Professor, Principal Investigator — Sun yat-sen universtiy cancer center
Locations (1):
- Sun yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Wang H, Wei J, Zheng Q, Meng L, Xin Y, Yin X, Jiang X. Radiation-induced heart disease: a review of classification, mechanism and prevention. Int J Biol Sci. 2019 Aug 8;15(10):2128-2138. doi: 10.7150/ijbs.35460. eCollection 2019. PMID 31592122
- [Background] Beukema JC, van Luijk P, Widder J, Langendijk JA, Muijs CT. Is cardiac toxicity a relevant issue in the radiation treatment of esophageal cancer? Radiother Oncol. 2015 Jan;114(1):85-90. doi: 10.1016/j.radonc.2014.11.037. Epub 2014 Dec 30. PMID 25554226
- [Background] Dess RT, Sun Y, Matuszak MM, Sun G, Soni PD, Bazzi L, Murthy VL, Hearn JWD, Kong FM, Kalemkerian GP, Hayman JA, Ten Haken RK, Lawrence TS, Schipper MJ, Jolly S. Cardiac Events After Radiation Therapy: Combined Analysis of Prospective Multicenter Trials for Locally Advanced Non-Small-Cell Lung Cancer. J Clin Oncol. 2017 May 1;35(13):1395-1402. doi: 10.1200/JCO.2016.71.6142. Epub 2017 Mar 16. PMID 28301264
- [Background] Atkins KM, Rawal B, Chaunzwa TL, Lamba N, Bitterman DS, Williams CL, Kozono DE, Baldini EH, Chen AB, Nguyen PL, D'Amico AV, Nohria A, Hoffmann U, Aerts HJWL, Mak RH. Cardiac Radiation Dose, Cardiac Disease, and Mortality in Patients With Lung Cancer. J Am Coll Cardiol. 2019 Jun 18;73(23):2976-2987. doi: 10.1016/j.jacc.2019.03.500. PMID 31196455
- [Background] Bradley JD, Paulus R, Komaki R, Masters G, Blumenschein G, Schild S, Bogart J, Hu C, Forster K, Magliocco A, Kavadi V, Garces YI, Narayan S, Iyengar P, Robinson C, Wynn RB, Koprowski C, Meng J, Beitler J, Gaur R, Curran W Jr, Choy H. Standard-dose versus high-dose conformal radiotherapy with concurrent and consolidation carboplatin plus paclitaxel with or without cetuximab for patients with stage IIIA or IIIB non-small-cell lung cancer (RTOG 0617): a randomised, two-by-two factorial phase 3 study. Lancet Oncol. 2015 Feb;16(2):187-99. doi: 10.1016/S1470-2045(14)71207-0. Epub 2015 Jan 16. PMID 25601342
- [Background] Wang K, Eblan MJ, Deal AM, Lipner M, Zagar TM, Wang Y, Mavroidis P, Lee CB, Jensen BC, Rosenman JG, Socinski MA, Stinchcombe TE, Marks LB. Cardiac Toxicity After Radiotherapy for Stage III Non-Small-Cell Lung Cancer: Pooled Analysis of Dose-Escalation Trials Delivering 70 to 90 Gy. J Clin Oncol. 2017 May 1;35(13):1387-1394. doi: 10.1200/JCO.2016.70.0229. Epub 2017 Jan 23. PMID 28113017
- [Background] Boekel NB, Schaapveld M, Gietema JA, Russell NS, Poortmans P, Theuws JC, Schinagl DA, Rietveld DH, Versteegh MI, Visser O, Rutgers EJ, Aleman BM, van Leeuwen FE. Cardiovascular Disease Risk in a Large, Population-Based Cohort of Breast Cancer Survivors. Int J Radiat Oncol Biol Phys. 2016 Apr 1;94(5):1061-72. doi: 10.1016/j.ijrobp.2015.11.040. Epub 2015 Dec 14. PMID 27026313
- [Background] Boero IJ, Paravati AJ, Triplett DP, Hwang L, Matsuno RK, Gillespie EF, Yashar CM, Moiseenko V, Einck JP, Mell LK, Parikh SA, Murphy JD. Modern Radiation Therapy and Cardiac Outcomes in Breast Cancer. Int J Radiat Oncol Biol Phys. 2016 Mar 15;94(4):700-8. doi: 10.1016/j.ijrobp.2015.12.018. Epub 2015 Dec 17. PMID 26972642
- [Background] Thatcher N, Hirsch FR, Luft AV, Szczesna A, Ciuleanu TE, Dediu M, Ramlau R, Galiulin RK, Balint B, Losonczy G, Kazarnowicz A, Park K, Schumann C, Reck M, Depenbrock H, Nanda S, Kruljac-Letunic A, Kurek R, Paz-Ares L, Socinski MA; SQUIRE Investigators. Necitumumab plus gemcitabine and cisplatin versus gemcitabine and cisplatin alone as first-line therapy in patients with stage IV squamous non-small-cell lung cancer (SQUIRE): an open-label, randomised, controlled phase 3 trial. Lancet Oncol. 2015 Jul;16(7):763-74. doi: 10.1016/S1470-2045(15)00021-2. Epub 2015 Jun 1. PMID 26045340
- [Background] Fossella FV, Lee JS, Murphy WK, Lippman SM, Calayag M, Pang A, Chasen M, Shin DM, Glisson B, Benner S, et al. Phase II study of docetaxel for recurrent or metastatic non-small-cell lung cancer. J Clin Oncol. 1994 Jun;12(6):1238-44. doi: 10.1200/JCO.1994.12.6.1238. PMID 7911160
- [Background] Kido H, Morizane C, Tamura T, Hagihara A, Kondo S, Ueno H, Okusaka T. Gemcitabine-induced pleuropericardial effusion in a patient with pancreatic cancer. Jpn J Clin Oncol. 2012 Sep;42(9):845-50. doi: 10.1093/jjco/hys099. Epub 2012 Jul 10. PMID 22782959
- [Background] Eremina V, Jefferson JA, Kowalewska J, Hochster H, Haas M, Weisstuch J, Richardson C, Kopp JB, Kabir MG, Backx PH, Gerber HP, Ferrara N, Barisoni L, Alpers CE, Quaggin SE. VEGF inhibition and renal thrombotic microangiopathy. N Engl J Med. 2008 Mar 13;358(11):1129-36. doi: 10.1056/NEJMoa0707330. PMID 18337603
- [Background] Wang J, Okazaki IM, Yoshida T, Chikuma S, Kato Y, Nakaki F, Hiai H, Honjo T, Okazaki T. PD-1 deficiency results in the development of fatal myocarditis in MRL mice. Int Immunol. 2010 Jun;22(6):443-52. doi: 10.1093/intimm/dxq026. Epub 2010 Apr 21. PMID 20410257
- [Background] Heinzerling L, Ott PA, Hodi FS, Husain AN, Tajmir-Riahi A, Tawbi H, Pauschinger M, Gajewski TF, Lipson EJ, Luke JJ. Cardiotoxicity associated with CTLA4 and PD1 blocking immunotherapy. J Immunother Cancer. 2016 Aug 16;4:50. doi: 10.1186/s40425-016-0152-y. eCollection 2016. PMID 27532025
- [Background] Brahmer J, Reckamp KL, Baas P, Crino L, Eberhardt WE, Poddubskaya E, Antonia S, Pluzanski A, Vokes EE, Holgado E, Waterhouse D, Ready N, Gainor J, Aren Frontera O, Havel L, Steins M, Garassino MC, Aerts JG, Domine M, Paz-Ares L, Reck M, Baudelet C, Harbison CT, Lestini B, Spigel DR. Nivolumab versus Docetaxel in Advanced Squamous-Cell Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Jul 9;373(2):123-35. doi: 10.1056/NEJMoa1504627. Epub 2015 May 31. PMID 26028407
- [Background] Curigliano G, Cardinale D, Dent S, Criscitiello C, Aseyev O, Lenihan D, Cipolla CM. Cardiotoxicity of anticancer treatments: Epidemiology, detection, and management. CA Cancer J Clin. 2016 Jul;66(4):309-25. doi: 10.3322/caac.21341. Epub 2016 Feb 26. PMID 26919165
- [Background] Ananthan K, Lyon AR. The Role of Biomarkers in Cardio-Oncology. J Cardiovasc Transl Res. 2020 Jun;13(3):431-450. doi: 10.1007/s12265-020-10042-3. Epub 2020 Jul 8. PMID 32642841
- [Background] Thavendiranathan P, Poulin F, Lim KD, Plana JC, Woo A, Marwick TH. Use of myocardial strain imaging by echocardiography for the early detection of cardiotoxicity in patients during and after cancer chemotherapy: a systematic review. J Am Coll Cardiol. 2014 Jul 1;63(25 Pt A):2751-68. doi: 10.1016/j.jacc.2014.01.073. Epub 2014 Apr 2. PMID 24703918
- [Background] Cardinale D, Colombo A, Bacchiani G, Tedeschi I, Meroni CA, Veglia F, Civelli M, Lamantia G, Colombo N, Curigliano G, Fiorentini C, Cipolla CM. Early detection of anthracycline cardiotoxicity and improvement with heart failure therapy. Circulation. 2015 Jun 2;131(22):1981-8. doi: 10.1161/CIRCULATIONAHA.114.013777. Epub 2015 May 6. PMID 25948538
- [Background] Malfatto G, Blengino S, Perego GB, Branzi G, Villani A, Facchini M, Parati G. Transthoracic impedance accurately estimates pulmonary wedge pressure in patients with decompensated chronic heart failure. Congest Heart Fail. 2012 Jan-Feb;18(1):25-31. doi: 10.1111/j.1751-7133.2011.00248.x. Epub 2011 Sep 14. PMID 22277174
- [Background] Parashar R, Bajpai M, Goyal M, Singh S, Tiwari S, Narayan VS. Impedance cardiography for monitoring changes in cardiac output. Indian J Physiol Pharmacol. 2012 Apr-Jun;56(2):117-24. PMID 23387239
- [Background] Siedlecka J, Siedlecki P, Bortkiewicz A. Impedance cardiography - Old method, new opportunities. Part I. Clinical applications. Int J Occup Med Environ Health. 2015;28(1):27-33. doi: 10.13075/ijomeh.1896.00451. PMID 26159944
- [Background] Lang CC, Agostoni P, Mancini DM. Prognostic significance and measurement of exercise-derived hemodynamic variables in patients with heart failure. J Card Fail. 2007 Oct;13(8):672-9. doi: 10.1016/j.cardfail.2007.05.004. PMID 17923361
- [Background] Lang CC, Karlin P, Haythe J, Lim TK, Mancini DM. Peak cardiac power output, measured noninvasively, is a powerful predictor of outcome in chronic heart failure. Circ Heart Fail. 2009 Jan;2(1):33-8. doi: 10.1161/CIRCHEARTFAILURE.108.798611. PMID 19808313